CLINICAL TRIAL: NCT07296016
Title: The Asia-Pacific Mitral & Tricuspid Valve-in-Valve/Valve-in-Ring Registry
Acronym: AP ViV
Status: Not yet recruiting | Type: Observational
Sponsor: Prince of Wales Hospital, Shatin, Hong Kong (Other)
Collaborators: National Heart Centre Singapore (Other)
Responsible Party: Principal Investigator, Dr So Chak Yu kent, Clinical Assistant Professor, Prince of Wales Hospital, Shatin, Hong Kong
Other Study IDs: 2025.502
Record Dates: First submitted 2025-11-21; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Structural Heart Disease; Mitral Valve Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prospective: Patient planned to undergo a Mitral valve-in-valve/valve-in-ring procedure.
- Retrospective: Patient that had at least one documented Mitral valve-in-valve/valve-in-ring procedure done during the period of 1 Jan 2023 to current date.

SUMMARY:
A significant number of patients with severe mitral and tricuspid valve disease have been previously treated with either valve repair with annuloplasty rings or valve replacement with bioprosthetic/mechanical valves. Over time, these bioprosthetic valves and rings may fail resulting in recurrence of the valvular disease. The technical aspects of a re-do operation are complex and these patients are often times at high risk for repeat open surgery. The emergence of transcatheter options may provide a safer and less invasive alternative to open surgery. Majority of the data currently exist for Western cohorts with limited longer-term outcomes. Data on this therapy is particularly lacking in the Asia-Pacific region, especially important in the light of known differences in body habitus and size.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 21
2. Had at least one documented Mitral valve-in-valve/valve-in-ring procedure done during the period of 1 Jan 2023 to current date. (Retrospective) OR Planned to undergo a Mitral valve-in-valve/valve-in-ring procedure. (Prospective) OR Had at least one documented Tricuspid valve-in-valve/valve-in-ring procedure done during the period of 1 Jan 2023 to current date. (Retrospective) OR Planned to undergo a Tricuspid valve-in-valve/valve-in-ring procedure. (Prospective)

Exclusion Criteria:

1. Active endocarditis
2. Any other conditions which investigator deems unsuitable for participation.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a retrospective and prospective, observational, multicenter cohort study of consecutive patients undergoing transcatheter mitral/tricuspid ViV or ViR procedure with balloon expandable valve across participating sites in Asia-Pacific from 1 Jan 2023 to 31 Dec 2035.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2035-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 10 years
  Rate of All-cause mortality in enrolled patients

SECONDARY OUTCOMES:
Procedural technical success rate | Immediately after operation
  Rate of Procedural technical success (defined per Mitral Valve Academic Research Consortium (MVARC) criteria at exit from the hybrid suite as patient alive with successful access, delivery, and retrieval of the device delivery system, successful deployment and correct position of the first intended device, and freedom from emergency surgery or reintervention associated with the device or access procedure)
Procedural complication rate | Periprocedural
  Rate of Procedural technical success (defined per Mitral Valve Academic Research Consortium (MVARC) criteria at exit from the hybrid suite as patient alive with successful access, delivery, and retrieval of the device delivery system, successful deployment and correct position of the first intended device, and freedom from emergency surgery or reintervention associated with the device or access procedure)
Major adverse cardiovascular events rate | 10 years
  Rate of Major adverse cardiovascular events in enrolled patients
New York Heart Association (NYHA) classification | 10 years
  NYHA class of enrolled patients
Echocardiographic result | 10 years
  Rate of Major adverse cardiovascular events in enrolled patients

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No